CLINICAL TRIAL: NCT02817919
Title: Modified Cohort Event Monitoring Of Injectable Artesunate, Artemether And Quinine In Ethiopia, Ghana, Malawi And Uganda
Brief Title: Cohort Event Monitoring in Sub Saharan Africa
Acronym: CEMISA
Status: Completed | Type: Observational
Sponsor: African Collaborating Centre for Pharmacovigilance (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: PV001
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2016-06

CONDITIONS: Malaria
Keywords: Pharmacovigilance; Africa
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This cohort event monitoring will document real-life safety experiences following the intake of Injectable AS. Specifically, the study will record common adverse events that are associated with the use of Inj. AS and associating factors such as age and gender that make some of these events more likely. The sample size of 3000 patients will enable the documentation of causally-related events that occur at frequencies of 1 in 1000 or more. Since quinine, the previous gold standard for treating severe malaria may still be used by facilities in addition to artesunate and artemether, the study will concurrently monitor the safety of these products though focus of the study is the capture of adverse events following exposure to Inj. AS. The concurrent monitoring of both quinine and artemether will also enable treatment practices in the study areas to be documented.

DETAILED DESCRIPTION:
Malaria is a preventable and treatable disease caused by Plasmodium species. In 2015, It was estimated that, about 1.8 million cases of malaria and about 400, 000 deaths were reported, 90% of which are in Africa. Those children who do not die may suffer brain damage or experience cognitive and learning deficits as a result of the disease severity. Though significant progress has been made in the last decade towards achieving global malaria targets, the disease burden is still relatively high in sub-Saharan African countries, especially among children <5 years of age.

Injectable artesunate (Inj. AS) is a life-saving medication indicated for the treatment of severe/complicated malaria either intravenously or intramuscularly. The current version (3rd edition) of the World Health Organization (WHO) Guidelines for the Treatment of Malaria strongly recommends, based on high-quality evidence, that adults and children with severe malaria should be treated with "intravenous or intramuscular artesunate". Injectable Artesunate is prequalified under the WHO Prequalification Scheme. It has received marketing authorization in nearly all malaria-endemic countries and millions of doses have been distributed for use in the management of severe malaria.

Despite the widespread usage of Inj. AS, the safety database for the product is nearly empty with the WHO Individual Case Safety Reports (ICSR) database containing only 2622 reports to artesunate including Inj AS. Inj AS is considered a safe product even though there have been reports of rare but serious haematological reactions in relation to its use including post-treatment haemolysis and subsequent anaemia, some of them life-threatening and requiring blood transfusion. Experts agree that the benefits of Inj. AS far outweigh any risks it may pose and this formed the basis for the WHO recommendation for the use of Inj. AS as the first product of choice for treating severe malaria except where it is not available and in which case parenteral artemether is recommended conditionally. In view of the millions of doses of Inj AS deployed and used each year, it is important to undertake focused, intensive safety surveillance of the medicine to obtain continuous evidence on its benefits-risk profile and also to prevent undocumented or rare but serious adverse events acting as barriers to its uptake.

Apart from the detailed well-collected safety information obtained during clinical trials, there is no published information on the real-life safety experience of Inj. AS in large cohorts of patients. This study is therefore designed to obtain real-life safety experience of Inj. AS when used in actual practice settings in 4 African countries - Ethiopia, Ghana, Malawi and Uganda. The study is designed as a prospective, observational, longitudinal cohort study of patients administered Inj AS in the course of normal clinical practice. The method used is cohort event monitoring which has been deployed for the study of antimalarials and is being suggested as a key method for several post-authorisation safety studies

ELIGIBILITY:
Inclusion criteria

* Severe Malaria (Plasmodia of any species) diagnosed as per national policies and health facility practice/protocol
* Ability and willingness to participate by giving signed informed consent. In the case of some adults and all children, signed informed consent would be obtained from the patient or a carer/guardian.
* Participants who agree to for follow-up visits and can be contacted by phone.

Exclusion criteria

* Patients (or carers/guardians) unwilling or unable to provide signed informed consent
* Patients with any illness that the investigator feels would be harmful to them to participate in the study
* Has not received Inj AS, AR, or Q.
* Existence of serious concurrent illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are diagnosed as having severe malaria.
Sampling Method: Non-Probability Sample
Enrollment: 1126 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The proportion of adverse events following administration of Injectable artesunate. | 28 days after administration of injectable artesunate

SECONDARY OUTCOMES:
The proportion of adverse events following administration of injectable artemether (AR) or Injectable quinine (Q) | 28 days after administration of injectable artemether or injectable quinine
The proportion of severe malaria cases that are treated with injectable. artesunate, artemether or quinine. | through study completion, an average of 1 year
Availability and stock levels of injectable artesunate, artemether or quinine in participating health facilities. | through study completion, an average of 1 year

OTHER OUTCOMES:
The proportion of treatment adherence to national treatment guidelines for severe malaria management. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kwaku P. Asante, MD, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana; Alexander NO Dodoo, PhD, Principal Investigator — WHO Collaborating Centre for Advocacy and Training in Pharmacovigilance
Locations (4):
- Ghana (4):
  - Kintampo North Municipal Hospital, Kintampo, Brong Ahafo Region
  - Princess Marie Louise Children's Hospital, Accra, Greater Accra Region
  - Ridge Hospital, Accra, Greater Accra Region
  - Agogo Presbytarian Hospital, Agogo

REFERENCES:
- [Derived] Ampadu HH, Dodoo ANO, Bosomprah S, Akakpo S, Hugo P, Gardarsdottir H, Leufkens HGM, Kajungu D, Asante KP. Safety Experience During Real-World Use of Injectable Artesunate in Public Health Facilities in Ghana and Uganda: Outcomes of a Modified Cohort Event Monitoring Study (CEMISA). Drug Saf. 2018 Sep;41(9):871-880. doi: 10.1007/s40264-018-0667-x. PMID 29696507